CLINICAL TRIAL: NCT04302922
Title: An Observational Study on the Association Between the Individual Chronotype and Body Composition Among German Students Aged 18 to 25 Years- The ChroNu Cohort
Brief Title: Association Between the Individual Chronotype and Body Composition in German Students - The ChroNu Study
Acronym: ChroNuCohort
Status: Completed | Type: Observational
Sponsor: Paderborn University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Anette Buyken, Prof. Dr. Anette Buyken, Public Health Nutrition, Paderborn University
Other Study IDs: BU 1807/3-2
Record Dates: First submitted 2020-01-22; First posted 2020-03-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Chronotype; social jetlag; body composition; meal timing; timing of physical activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronotype is defined as the midpoint of sleep and describes a biological construct of an organism's temporal organisation. Misalignment between the individual chronotype and socially determined schedules may result in a phenomenon called "social jetlag". Emerging evidence indicates that both, a later chronotype and/or a substantial "social jetlag" adversely affects metabolic health. Young adults may be particularly vulnerable to these exposures since the chronotype progressively delays from adolescence until early adulthood (approx. 20 years of age) before it advances again. Simultaneously, education in institutions or working hours starts early during the day, potentially contribute to substantial "social jetlag". Data on the development of overweight / obesity prevalence in Germany indicates that rates are now constant or declining in most adult age groups, with the clear exception of young adults, in whom rates continue to be on the rise. Nonetheless, the potential contribution of chronotype and/or social jetlag to this secular trend has not been addressed in Germany. Hence, the hypothesis of the ChroNu cohort is that individual chronotype and social jetlag are predictors of (changes in) the body composition in young adulthood (ages 18-25 years) and that changes in chronotype / social jetlag will result in changes in body composition. The ChroNu cohort forms part of the overall ChroNu study, which addresses the hypothesis that timing of food intake which diverges from the individual chronotype constitutes a characteristic of social jetlag which has adverse short- and long-term consequences for metabolic health (see The ChroNustudy). This study will recruit 300 healthy, non-obese students aged 18-25 years enrolled at Paderborn University until February 2020 and follow these up one year later. Chronotype and social jetlag will be determined using the validated MCTQ. Body composition will be assessed by bioimpedance analysis (BIA) The ChroNu cohort study will reveal important information on the relevance of a biologically determined phenomenon, i.e. the chronotype and the potentially resultant social jetlag for body composition development in a population vulnerable to increases in body fat.

DETAILED DESCRIPTION:
Background:

The chronotype is defined as the midpoint of sleep and describes biological construct of an organisms temporal organisation. It is itself determined by genetics, age, sex, and environment. Misalignment between the individual chronotype and socially determined schedules may result in a phenomenon which has been called "social jetlag". Emerging evidence indicates that a later chronotype and/or "social jetlag" predisposes to weight gain, higher BMI and higher odds for type 2 diabetes. A later chronotype has been also associated with a more adverse body composition. Since the chronotype progressively delays from adolescence until early adulthood (approx. 20 years of age), before it advances again, young adults may be particularly vulnerable to such adverse exposures. These exposures may result of a higher evening energy intake which in turn was observed for a later chronotype at adolescence. A preferred consumption of energy intake in the evening lead to higher total energy intake. Social schedules such as early starting hours at schools and universities, which potentially contribute to substantial "social jetlag", may influence individual meal timing. The chronotype, however, may be the main predictor for meal timing like skipping breakfast or not. However, it is not clear yet whether this affects predominantly early or late chronotypes in young adults.

Data on the development of overweight / obesity prevalence in Germany indicates that rates are now constant or declining in most adult age groups, with the clear exception of young adults, in whom rates continue to be on the rise. Nonetheless, the potential contribution of chronotype and/or social jetlag to this secular trend has not been addressed in Germany.

Hypothesis:

The hypothesis of the ChroNu cohort is that individual chronotype and social jetlag are predictors of (changes in) body composition in young adulthood (ages 18-25 years) and that changes in chronotype / social jetlag will result in changes in body composition.

Aim:

Hence, the investigators aim to study the association between the body composition and the chronotype / social jetlag at first stage and in a follow-up after one year the causal relationship between changes in chronotype/social jetlag and body composition.

Methods 1: participants In the ChroNu cohort study, the investigators will recruit at least 300 students from Paderborn University aged 18 -25 years. Students will be contacted via social media, mailing-lists, poster and flyer, and presentation of the study in lectures. The ChroNu cohort study will last from Sept 2019 to approximately Febr 2020. Due to the restrictions caused by the SARS-CoV2 pandemic, participants were recruited again in June 2020 to fill in an online survey consisting of the same questionairies as at baselineThe follow-up is scheduled for May - June 2022.

Methods 2: Methods:

In the screening of participants for ChroNu cohort study, eligible participants are asked to fill in the Munich Chronotype Questionnaire (MCTQ, © Roenneberg & co-workers 2015), which is a validated questionnaire to calculate the individual chronotype. In this questionnaire, participants are asked about their sleep timing separately for work days and work-free days: when they go to bed (bed time); when they prepare to sleep); how long it takes them to fall asleep (sleep latency); when they wake up (sleep end); and how long it takes them to get out of bed (sleep inertia). The mid-sleep point, which defines the chronotype, is calculated as the time when falling asleep plus half of the sleep duration. If the sleep duration is longer on free days than on work days this oversleep is corrected (corrected mid-sleep point): half of the difference in sleep duration is subtracted. Social jet lag is calculated as the difference between the mid-sleep time on work days and work-free days.

The individual body composition, which is the outcome of this study, is analyzed using Bioimpedance Analysis (BIA) (mBCA 515, SECA). For the analyses, waist circumference, body size and body weight are required: waist circumference is measured midway between the lowest rib and the iliac crest by trained personal following the World Health Organisation (WHO) recommendations and entered in the BIA device. Body size is measured by means of an ultrasonic measuring station (seca 287 dp) from SECA and directly transferred to the BIA device. For measurement of body weight and body composition participants need to stand on the BIA device.

Since the chronotype and potentially resultant social jetlag is affected by environment, participants are asked to fill in additional questionnaires on their daily routines and diurnal patterns in both physical activity and meal timing and food intake. Questions on daily routine include start and end time of both university and work if applicable.

For a following ChroNu nutritional trial, the investigators are looking for the earliest and latest chronotypes among our ChoNu cohort. Participants each with the earliest and the latest mid-sleep points among our cohort seem to be suitable.

Statistical analyses Linear mixed-effects regression models are used to analyze the associations between chronotype (continuously in h:mm) as predictor and BMI, body fat, and visceral fat. The same analyses will be performed for social jetlag as predictor.

Multivariable linear and logistic mixed-effects regression models are performed to investigate associations between the chronotype and the circadian patterns of meal timing and physical activity. In second step, multivariable regression analysis is used to examine if the assocation between chronotype and body composition is mediated by the circadian patterns of both meal timing and physical activity. All basic models will be adjusted for age and additionally adjusted for potentially confounders which were considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy students of Paderborn University
* 18-25 years old

Exclusion Criteria:

* Students studying nutrition science
* shift work in the past 3 months
* crossing of >1 time zone in the past 3 months
* pregnancy
* lactation
* intake of medication such as antidepressants or sleeping pills

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: students of Paderborn University (see inclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change of body fat content from pre-post Covid-19 pandemic | Body fat will be measured both at baseline after enrolment and post-pandemic (follow up).
  Body fat content [kg] is measured by bio-impedance analysis (BIA)

SECONDARY OUTCOMES:
Change in weight from pre-post Covid-19 pandemic | Anthropometric measurements (weight, height, waist circumference) will be performed together with the BIA measurements both at baseline and post-pandemic (follow-up) and are expected to last approximately 20 minutes each.
  Body weight is measured in kilograms simultaneously when participants are measured for body composition on the BIA device.
Change in height from pre-post Covid-19 pandemic | Anthropometric measurements (weight, height, waist circumference) will be performed together with the BIA measurements both at baseline and post-pandemic (follow-up) and are expected to last approximately 20 minutes each.
  Body height is measured in meters simultaneously when participants are measured for body composition on the BIA device.
Change in BMI from pre-post Covid-19 pandemic | Anthropometric measurements (weight, height, waist circumference) will be performed together with the BIA measurements both at baseline and post-pandemic (follow-up) and are expected to last approximately 20 minutes each.
  Weight and height will be combined to report BMI in kg/m^2
Change in waist circumference from pre-post Covid-19 pandemic | Anthropometric measurements (weight, height, waist circumference) will be performed together with the BIA measurements both at baseline and post-pandemic (follow-up) and are expected to last approximately 20 minutes each.
  Waist circumference is measured midway between the lowest rib and the iliac crest in centimeters.
Change in daily routine and physical activity from pre-post Covid-19 pandemic | The questionaires concerning daily routine, physical activity, meal timing and food frequency will be performed at baseline and post-pandemic (follow-up) and are expected to last approximately 45 minutes each.
  Participants are asked to fill in additional questionnaires on diurnal patterns of physical activity. The scale is the frequency of physical activity with the maximum value being "every day" and the minimum value being "never". All questionnaires are based on the last 4 weeks comparable to the time frame to calculate the chronotype.
Change in meal timing from pre-post Covid-19 pandemic | The questionaires concerning daily routine, physical activity, meal timing and food frequency will be performed at baseline and post-pandemic (follow-up) and are expected to last approximately 45 minutes each.
  Participants are asked to fill in additional questionnaires on diurnal patterns of meal timing. Participants are asked to select between breakfast, lunch, dinner and snack times on each day. All questionnaires are based on the last 4 weeks comparable to the time frame to calculate the chronotype.
Change in food choice from pre-post Covid-19 pandemic | The questionaires concerning daily routine, physical activity, meal timing and food frequency will be performed at baseline and post-pandemic (follow-up) and are expected to last approximately 45 minutes each.
  Food choice: Participants are asked to fill in additional questionnaires on food intake. Food intake is obtained using a food frequency questionnaire. Questions on beverages are based on the validated German food frequency questionaires (FFQ) "Studie zur Gesundheit Erwachsener in Deutschland" (DEGS). Food intake is based on FFQ, which has not been validated yet, additional to DEGS. Only those questions were selected that ask about the food frequency of different carbohydrate sources. All questionnaires are based on the last 4 weeks comparable to the time frame to calculate the chronotype.

CONTACTS AND LOCATIONS:
Overall Officials: Anette E Buyken, Prof. Dr., Principal Investigator — Paderborn University
Locations (1):
- Paderborn University, Paderborn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.